CLINICAL TRIAL: NCT04231201
Title: Aortic Stenosis: Evaluation of Severity Before and After Transcatheter Aortic Valve Implantation by Means of Ballistocardiography and Seismocardiography.
Brief Title: Aortic Stenosis Evaluated Via Modern Ballistocardiography and Seismocardiography
Acronym: TAVI
Status: Suspended | Type: Observational
Why Stopped: COVID pandemic
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2019/596
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Aortic Stenosis
Keywords: Ballistocariodgraphy; Seismocardiography; LV mechanics
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Calcific aortic stenosis (AS) (formerly "senile" or "degenerative") is a frequent disease of heart valves and is characterized by a thickness and calcification of leaflets with a significant increase of the pressure gradient, defined as an aortic jet velocity of > 2 m/s. Whenever the aortic jet velocity is > 4 m/s, in association with an aortic valve area of < 1 cm2, the disease is classified as severe and cardiac outflow obstruction develops. AS affects 1-2% of population aged of > 65 years and 12% of those aged > 75 years. Among those aged > 75 years, it is estimated that 3.5% has severe AS. With the aging of population, the prevalence of AS is expected to increase in the forthcoming years. Transcatheter Aortic Valve Implantation (TAVI) has been introduced in 2004 and consists in percutaneous replacement of the aortic valve. It is indicated in those patients with severe AS who cannot undergo surgical replacement because of high surgical risk. TAVI seems to be a good alternative to surgical intervention also for patients deemed at intermediate risk, especially if they are frail or aged. Ballistocardiography (BCG) consists of the measurement of the body's accelerations as a consequence of the recoil forces generated by the blood mass ejection at each cardiac contraction and recorded on the body's surface close to the subject's center of mass. Seismocardiography (SCG) records the heart-induced accelerations generated at each cardiac contraction and transmitted to the local chest surface. Thanks to specific algorithms applied to the SCG and BCG waves, it is possible to compute the kinetic energy (KE) and Power (P) of a single cardiac contractile cycle.

The aims of our study are to demonstrate that: LVOT Vmax and LVOT VTI changes obtained with echocardiography can be estimated reliably throught BCG and SCG signals, before and after TAVI procedure; Pmax and KE computed from the BCG and SCG signals could predict the severity of the AS before the TAVI procedure.

KE and P computed from non invasively recorded BCG and SCG waves may prove useful in the evaluation of AS severity and its evolution before and after TAVI procedure, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Severe aortic stenosis, planned to undergo TAVI procedure

Exclusion Criteria:

* Concomitant heart valve disease other than AS
* C2 and D2 stages of AS according to the current definition (see table I for further details)
* Heart failure regardless to the etiology
* Arrhythmias
* Severe kidney disease
* Denied consent to participate

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient population studied: patients with aortic stenosis planned to undergo TAVI procedure.
  Number of patients planned: since this is a pilot study, no formal simple size calculation can be done. The Cardiology department of the Erasme hospital perform an average of 3 TAVI procedure a month. Since the enrollment will take place from January to September 2023, a total of 135 patients will be enrolled. Because of a complication rate of 10% linked to the invasive procedure, we expect 100 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of cardiac kinetic energy before and after aortic valve replacement by the means of modern micro-accelerometers and gyroscopes, namely ballistocardiography (BCG) and seismocardiography (SCG). | 3 years
  Kinetic energy (1/2 mv^2, J) and its temporal integral are computed from the BCG and SCG signals before and after valvular replacement.
Measurement of cardiac Power before and after aortic valve replacement by the means of modern micro-accelerometers and gyroscopes, namely ballistocardiography (BCG) and seismocardiography (SCG). | 3 years
  Maximal power (F*v, J/s)* produced during a contractile cycle is computed from the BCG and SCG signals before and after valvular replacement.
  * F= Force (mass*acceleration) (Kg*m/s^2) v= velocity (m/s)

SECONDARY OUTCOMES:
Measurement of LV twist and global longitudinal strain before and after valvular replacement | 3 years
  From 2 dimensional speckle tracking imaging (2D-STI) echocardiography, LV twist (°) and global longitudinal strain (°) will be measured before and after valvular replacement

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Morra, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided